CLINICAL TRIAL: NCT04551963
Title: A Drug-Drug Interaction Study of Zanubrutinib With Moderate and Strong CYP3A Inhibitors in Patients With B-Cell Malignancies
Brief Title: Interaction Study of Zanubrutinib With Moderate and Strong CYP3A Inhibitors in Participants With B-Cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-113
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2023-11-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: B-cell Malignancies
MeSH Terms: interventions — zanubrutinib; Fluconazole; Diltiazem; Voriconazole; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Zanubrutinib with or without Moderate CYP3A (Experimental): Cycle 1 (30 days): Participants were administered zanubrutinib at a dose of 320 mg once a day from Day 1 to Day 3; From Day 4 to Day 10, fluconazole was administered once a day at a dose of 400 mg with zanubrutinib at a reduced dose of 80 mg twice a day; On Day 11 and Day 12, zanubrutinib monotherapy was administered at 80 mg twice a day, followed by 320 mg once a day from Day 13 to Day 21; From Day 22 to Day 28, diltiazem was administered once a day at a dose of 180 mg with 80 mg zanubrutinib twice a day; On Day 29 and Day 30, zanubrutinib monotherapy was administered 80 mg twice a day.
  Cycles 2 to 6 (28 days each cycle): Zanubrutinib 160 mg twice a day or 320 mg once a day.
  Interventions: Drug: Zanubrutinib; Drug: Fluconazole; Drug: Diltiazem
- Arm B: Zanubrutinib with or without Strong CYP3A (Experimental): Cycle 1 (30 days): Participants were administered zanubrutinib at a dose of 320 mg once a day from Day 1 to Day 3; From Day 4 to Day 10, voriconazole was administered twice a day at a dose of 200 mg (total daily dose of 400 mg) with zanubrutinib at a reduced dose of 80 mg once a day; On Day 11 and Day 12, zanubrutinib monotherapy was administered at 80 mg once a day, followed by 320 mg once a day from Day 13 to Day 21; From Day 22 to Day 28, clarithromycin was administered twice a day at a dose of 250 mg (total daily dose of 500 mg) with 80 mg zanubrutinib once a day; On Day 29 and Day 30, zanubrutinib monotherapy was administered 80 mg once a day.
  Cycles 2 to 6 (28 days each cycle): Zanubrutinib 160 mg twice a day or 320 mg once a day.
  Interventions: Drug: Zanubrutinib; Drug: Voriconazole; Drug: Clarithromycin

INTERVENTIONS:
Drug: Zanubrutinib — Capsules administered at a dose and frequency as specified in the treatment arm
  Other Names: BGB-3111; BRUKINSA
Drug: Fluconazole — Capsules administered at a dose and frequency as specified in the treatment arm
  Arms: Arm A: Zanubrutinib with or without Moderate CYP3A
Drug: Diltiazem — Capsules administered at a dose and frequency as specified in the treatment arm
  Arms: Arm A: Zanubrutinib with or without Moderate CYP3A
Drug: Voriconazole — Capsules administered at a dose and frequency as specified in the treatment arm
  Arms: Arm B: Zanubrutinib with or without Strong CYP3A
Drug: Clarithromycin — Capsules administered at a dose and frequency as specified in the treatment arm
  Arms: Arm B: Zanubrutinib with or without Strong CYP3A

SUMMARY:
The primary objective of this study was to assess the steady-state zanubrutinib pharmacokinetics (PK) when co-administered with moderate and strong cytochrome P450 family 3 subfamily A (CYP3A) inhibitors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed CLL/SLL, MCL, WM, or MZL.
2. Relapsed or refractory disease after at least 1 prior line of systemic therapy. Participants with MZL are required to have failed an anti-CD20 monoclonal antibody-containing chemotherapy regimen.
3. Baseline Eastern Cooperative Oncology Group performance status of 0 to 1.
4. Meet protocol guidelines for adequate bone marrow, kidney, liver, and cardiac function.

Key Exclusion Criteria:

1. Requirement of chronic treatment with strong and moderate CYP3A inhibitors or inducers or with drugs that are not allowed to be used in combination with diltiazem, clarithromycin, fluconazole, or voriconazole.
2. History of stroke or intracranial hemorrhage (within 6 months of treatment start).
3. Known hypersensitivity or contraindication to zanubrutinib, diltiazem, clarithromycin, fluconazole, or voriconazole.
4. Prior exposure to zanubrutinib or other Bruton tyrosine kinase inhibitor
5. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (7):
- Australia (7):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - John Flynn Private Hospital, Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford PK, South Australia
  - Monash Health, Clayton, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Tariq B, Ou YC, Stern JC, Mundra V, Wong Doo N, Walker P, Lewis KL, Lin C, Novotny W, Sahasranaman S, Opat S. A phase 1, open-label, randomized drug-drug interaction study of zanubrutinib with moderate or strong CYP3A inhibitors in patients with B-cell malignancies. Leuk Lymphoma. 2023 Feb;64(2):329-338. doi: 10.1080/10428194.2022.2150820. Epub 2022 Dec 8. PMID 36480811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 study centers in Australia.
Period: Overall Study
Arm/Group | Arm A: Zanubrutinib With or Without Moderate CYP3A | Arm B: Zanubrutinib With or Without Strong CYP3A
Started | 13 | 13
Completed | 11 | 12
Not Completed | 2 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Zanubrutinib With or Without Moderate CYP3A | Arm B: Zanubrutinib With or Without Strong CYP3A | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.5 (9.85) | 71.8 (8.64) | 71.1 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Arm A: Area Under Plasma Concentration-time Curve up to the Last Measurable Concentration (AUC0-t)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: The pharmacokinetic (PK) analysis set included all participants who received at last 1 dose of zanubrutinib and had evaluable PK data (at least 1 PK parameter could be calculated).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Arm A: Zanubrutinib With or Without Moderate CYP3A: Cycle 1 (30 days): Participants were administered zanubrutinib at a dose of 320 mg once a day (QD) from Day 1 to Day 3; From Day 4 to Day 10, fluconazole was administered once a day at a dose of 400 mg with zanubrutinib at a reduced dose of 80 mg twice a day (BID); On Day 11 and Day 12, zanubrutinib monotherapy was administered at 80 mg twice a day, followed by 320 mg once a day from Day 13 to Day 21; From Day 22 to Day 28, diltiazem was administered once a day at a dose of 180 mg with 80 mg zanubrutinib twice a day; On Day 29 and Day 30, zanubrutinib monotherapy was administered 80 mg twice a day.
  Cycles 2 to 6 (28 days each cycle): Zanubrutinib 160 mg twice a day or 320 mg once a day.
Arm/Group | Arm A: Zanubrutinib With or Without Moderate CYP3A
Number analyzed (Participants) | 13
h*ng/mL
  Zanubrutinib 320 mg QD | 1899.32 (44.95)
  Zanubrutinib 80 mg BID + 400 mg fluconazole QD | 921.63 (45.80)
  Zanubrutinib 80 mg BID + 180 mg diltiazem QD | 797.87 (43.05)
Statistical Analysis 1: Comparison: Arm A: Zanubrutinib With or Without Moderate CYP3A; Arm A: Zanubrutinib alone vs. Zanubrutinib + fluconazole; Test type: Equivalence — Two one sided tests procedure by estimation of ratio of geometric means and 90% CI; exponential transformation from estimated difference in natural logarithm scale obtained from linear mixed effect model with treatment as a fixed effect and participant as a random effect; Ratio of geometric least squares mean = 0.49, 90% CI 2-sided [0.42 to 0.56]
Statistical Analysis 2: Comparison: Arm A: Zanubrutinib With or Without Moderate CYP3A; Arm a: Zanubrutinib alone vs. Zanubrutinib + diltiazem; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.42, 90% CI 2-sided [0.34 to 0.51]

2. Primary Outcome: Arm B: Area Under Plasma Concentration-time Curve up to the Last Measurable Concentration (AUC0-t)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: The PK analysis set included all participants who received at last 1 dose of zanubrutinib and had evaluable PK data (at least 1 PK parameter could be calculated).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Arm B: Zanubrutinib With or Without Strong CYP3A: Cycle 1 (30 days): Participants were administered zanubrutinib at a dose of 320 mg once a day from Day 1 to Day 3; From Day 4 to Day 10, voriconazole was administered twice a day at a dose of 200 mg (total daily dose of 400 mg) with zanubrutinib at a reduced dose of 80 mg once a day; On Day 11 and Day 12, zanubrutinib monotherapy was administered at 80 mg once a day, followed by 320 mg once a day from Day 13 to Day 21; From Day 22 to Day 28, clarithromycin was administered twice a day at a dose of 250 mg (total daily dose of 500 mg) with 80 mg zanubrutinib once a day; On Day 29 and Day 30, zanubrutinib monotherapy was administered 80 mg once a day.
Arm/Group | Arm B: Zanubrutinib With or Without Strong CYP3A
Number analyzed (Participants) | 13
h*ng/mL
  Zanubrutinib 320 mg QD | 1550.40 (49.20)
  Zanubrutinib 80 mg QD + 200 mg voriconazole BID | 1254.29 (22.36)
  Zanubrutinib 80 mg QD + 250 mg clarithromycin BID | 763.00 (54.79)
Statistical Analysis 1: Comparison: Arm B: Zanubrutinib With or Without Strong CYP3A; Arm B: Zanubrutinib alone vs. zanubrutinib + voriconazole; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.81, 90% CI 2-sided [0.66 to 0.99]
Statistical Analysis 2: Comparison: Arm B: Zanubrutinib With or Without Strong CYP3A; Arm B: Zanubrutinib alone vs zanubrutinib + clarithromycin; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.49, 90% CI 2-sided [0.41 to 0.58]

3. Primary Outcome: Arm A: Area Under Plasma Concentration-time Curve From Time 0 Extrapolated to 24 Hours (AUC0-24h)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Arm A: Zanubrutinib With or Without Moderate CYP3A
Number analyzed (Participants) | 12
h*ng/mL
  Zanubrutinib 320 mg QD | 2035.32 (46.97)
  Zanubrutinib 80 mg BID + 400 mg fluconazole QD | 1911.93 (46.97)
  Zanubrutinib 80 mg BID + 180 mg diltiazem QD | 1653.07 (44.88)
Statistical Analysis 1: Comparison: Arm A: Zanubrutinib With or Without Moderate CYP3A; Arm A: Zanubrutinib alone vs. zanubrutinib + fluconazole; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.94, 90% CI 2-sided [0.82 to 1.08]
Statistical Analysis 2: Comparison: Arm A: Zanubrutinib With or Without Moderate CYP3A; Arm A: Zanubrutinib alone vs. zanubrutinib + diltiazem; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.81, 90% CI 2-sided [0.66 to 0.99]

4. Primary Outcome: Arm B: Area Under Plasma Concentration-time Curve From Time 0 Extrapolated to 24 Hours (AUC0-24h)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Arm B: Zanubrutinib With or Without Strong CYP3A
Number analyzed (Participants) | 12
h*ng/mL
  Zanubrutinib 320 mg QD | 1578.12 (49.53)
  Zanubrutinib 80 mg QD + 200 mg voriconazole BID | 1376.02 (25.09)
  Zanubrutinib 80 mg QD + 250 mg clarithromycin BID | 766.71 (60.44)
Statistical Analysis 1: Comparison: Arm B: Zanubrutinib With or Without Strong CYP3A; Arm B: Zanubrutinib alone vs. zanubrutinib + voriconazole; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.83, 90% CI 2-sided [0.65 to 1.06]
Statistical Analysis 2: Comparison: Arm B: Zanubrutinib With or Without Strong CYP3A; Arm B: Zanubrutinib alone vs zanubrutinib + clarithromycin; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.48, 90% CI 2-sided [0.40 to 0.58]

5. Primary Outcome: Arm A: Maximum Observed Concentration (Cmax)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm A: Zanubrutinib With or Without Moderate CYP3A
Number analyzed (Participants) | 13
ng/mL
  Zanubrutinib 320 mg QD | 520.78 (39.18)
  Zanubrutinib 80 mg BID + 400 mg fluconazole QD | 235.72 (42.53)
  Zanubrutinib 80 mg BID + 180 mg diltiazem QD | 211.06 (36.59)
Statistical Analysis 1: Comparison: Arm A: Zanubrutinib With or Without Moderate CYP3A; Arm A: Zanubrutinib alone vs. zanubrutinib + fluconazole; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.45, 90% CI 2-sided [0.35 to 0.58]
Statistical Analysis 2: Comparison: Arm A: Zanubrutinib With or Without Moderate CYP3A; Arm A: Zanubrutinib alone vs. zanubrutinib + diltiazem; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.41, 90% CI 2-sided [0.32 to 0.51]

6. Primary Outcome: Arm B: Maximum Observed Concentration (Cmax)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm B: Zanubrutinib With or Without Strong CYP3A
Number analyzed (Participants) | 13
ng/mL
  Zanubrutinib 320 mg QD | 428.88 (43.56)
  Zanubrutinib 80 mg QD + 200 mg voriconazole BID | 353.11 (30.23)
  Zanubrutinib 80 mg QD + 250 mg clarithromycin BID | 215.15 (51.79)
Statistical Analysis 1: Comparison: Arm B: Zanubrutinib With or Without Strong CYP3A; Arm B: Zanubrutinib alone vs. zanubrutinib + voriconazole; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.82, 90% CI 2-sided [0.68 to 1.00]
Statistical Analysis 2: Comparison: Arm B: Zanubrutinib With or Without Strong CYP3A; Arm B: Zanubrutinib alone vs. zanubrutinib + clarithromycin; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.50, 90% CI 2-sided [0.39 to 0.64]

7. Primary Outcome: Arm A: Time of the Maximum Observed Concentration (Tmax)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm A: Zanubrutinib With or Without Moderate CYP3A
Number analyzed (Participants) | 13
Hours
  Zanubrutinib 320 mg QD | 2.03 [1.0 to 4.0]
  Zanubrutinib 80 mg BID + 400 mg fluconazole QD | 2.93 [1.0 to 4.0]
  Zanubrutinib 80 mg BID + 180 mg diltiazem QD | 2.05 [1.0 to 4.2]

8. Primary Outcome: Arm B: Time of the Maximum Observed Concentration (Tmax)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm B: Zanubrutinib With or Without Strong CYP3A
Number analyzed (Participants) | 13
Hours
  Zanubrutinib 320 mg QD | 3.00 [1.0 to 4.0]
  Zanubrutinib 80 mg QD + 200 mg voriconazole BID | 2.05 [1.0 to 3.9]
  Zanubrutinib 80 mg QD + 250 mg clarithromycin BID | 2.08 [0.5 to 7.9]

9. Primary Outcome: Arm A: Apparent Terminal Elimination Half-life (t1/2)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | Arm A: Zanubrutinib With or Without Moderate CYP3A
Number analyzed (Participants) | 13
Hours
  Zanubrutinib 320 mg QD | 2.15 [1.4 to 4.5]
  Zanubrutinib 80 mg BID + 400 mg fluconazole QD | 2.10 [1.7 to 3.3]
  Zanubrutinib 80 mg BID + 180 mg diltiazem QD | 2.14 [1.4 to 4.0]

10. Primary Outcome: Arm B: Apparent Terminal Elimination Half-life (t1/2)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8 and 10 hours on Cycle 1 Day 3, Day 10, and Day 28 (30-day cycle)
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | Arm B: Zanubrutinib With or Without Strong CYP3A
Number analyzed (Participants) | 13
Hours
  Zanubrutinib 320 mg QD | 1.79 [1.2 to 2.5]
  Zanubrutinib 80 mg QD + 200 mg voriconazole BID | 2.38 [1.6 to 2.8]
  Zanubrutinib 80 mg QD + 250 mg clarithromycin BID | 2.08 [1.4 to 2.9]

11. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including clinical laboratory tests
Time Frame: From the date of first study drug administration to 30 days after last dose (up to approximately 15 months)
Population: The safety analysis set included all participants who were enrolled and received any dose of zanubrutinib
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Zanubrutinib With or Without Moderate CYP3A | Arm B: Zanubrutinib With or Without Strong CYP3A
Number analyzed (Participants) | 13 | 13
Participants
  At least one TEAE | 12 | 12
  At least one SAE | 3 | 1

ADVERSE EVENTS:
Time Frame: From the date of first study drug administration to 30 days after last dose (up to approximately 15 months)
Description: The safety analysis set included all participants who were enrolled and received any dose of zanubrutinib
Arm/Group | Arm A: Zanubrutinib With or Without Moderate CYP3A | Arm B: Zanubrutinib With or Without Strong CYP3A
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 3/13 | 1/13
Other Adverse Events (participants affected / at risk) | 12/13 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Zanubrutinib With or Without Moderate CYP3A (N=13) | Arm B: Zanubrutinib With or Without Strong CYP3A (N=13)
Fall (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Mantle cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Pneumonia cryptococcal (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Zanubrutinib With or Without Moderate CYP3A (N=13) | Arm B: Zanubrutinib With or Without Strong CYP3A (N=13)
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Fatigue (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT04551963/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT04551963/SAP_001.pdf